CLINICAL TRIAL: NCT04780750
Title: Phase III Study Comparing Concurrent Chemoradiotherapy With Weekly Docitaxel Plus Cisplatin Versus the Standard Concurrent Radiotherapy With Cisplatin in Patients With Locally Advanced Squamous Cell Carcinoma of the Head and Neck
Brief Title: Concurent Chemoradiotherapy in Head and Neck Cancers
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, doaa abd elaleem alsayed mohamed, principle investigator, Assiut University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: head and neck cancers
Record Dates: First submitted 2021-02-15; First posted 2021-03-03 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-02

CONDITIONS: Squamous Cell Carcinoma of Head and Neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Docetaxel

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A concurrent chemoradiotherapy with weekly docitaxel and cisplatin every 3 weeks (Active Comparator): Arm A (tested regimen): concurrent chemoradiotherapy with weekly docitaxel (20 mg\m2) and cisplatin (80mg\m2 every 3 weeks)
  Interventions: Drug: Docetaxel
- Arm B :concurrent chemoradiotherapy with cisplatin every 3 weeks (Active Comparator): Arm B (standard regimen):concurrent chemoradiotherapy with cisplatin (100mg\m2 every 3 weeks)
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: Docetaxel — Arm A (tested regimen): concurrent chemoradiotherapy with weekly docitaxel (20 mg\m2) and cisplatin (80mg\m2 every 3 weeks)
  Other Names: taxoter

SUMMARY:
To compare the efficacy and toxicities of the combination between weekly docitaxel and cisplatin (every3 week) concurrent with radiation versus the standard concurrent chemoradiotherapy with high dose cisplatin (100mg\m2) for locally advanced HNSCC

DETAILED DESCRIPTION:
Head and neck cancer is the eighth most common cancer in the United States . For locally advanced HNSCC, concurrent chemoradiotherapy (chemo-RT) is the standard treatment established with multiple randomized trials . The survival benefit of chemo-RT in locally advanced HNSCC has been confirmed by meta-analyses, which revealed a 19% reduction in mortality and an absolute survival benefit of 8% at 5years when chemotherapy was administered concurrently with radiation Despite incremental improvements in local regional control and survival in HNSCC patients treated with chemo-RT, a substantial fraction of patients suffer persistent or recurrent diseases. Combining novel agents with radiation therapy therefore remains of great interest to further improving the treatment outcomes of HNSCC .

Cisplatin is the most commonly used chemotherapeutic agent given concurrently with radiation. However, introduction of additional effective radiosensitizing agents is urgently needed. A significant percentage of patients appropriate for definitive concurrent chemo-RT are not candidates for cisplatin based treatment.

Furthermore, recent data have emerged that cisplatin might not be the most optimal cytotoxic radiosensitizing agent when addition of novel targeted agents to concurrent chemo-RT is evaluated.

Radiation Therapy Oncology Group (RTOG) 0234 is a phase II randomized clinical trial evaluating postoperative radiation plus concurrent docetaxel and cetuximab versus postoperative radiation plus cisplatin and cetuximab for high-risk HNSCC after surgery. The results showed an impressive improvement in overall survival and disease-free survival of the docetaxel arm compared to the cisplatin arm (79% versus 69% and 66% versus 57% respectively . These results are pointing to the possibility that a non-cisplatin based regimen chemo-RT should be explored for further development of novel targeted agents and led to a recently opened phase III randomized RTOG trial, RTOG 1216, which compares postoperative radiation with concurrent cisplatin versus docetaxel versus docetaxel and cetuximab for high-risk HNSCC patients . docetaxel appears to have active antitumor activity in advanced SCCHN . In preclinical studies, docetaxel leads to tumor cell reoxygenation and mitotic arrest with potent radiosensitization.

ELIGIBILITY:
Inclusion Criteria:

* pathologically confirmed squmous cell carcinoma performance status 0-1 adequte renal and hepatic function

Exclusion Criteria:

* poor performance status
* impaired renal or hepatic function

  =Squamous cell carcinoma of salivary gland,parotid and paranasal carcinomas were --0excluded from the study
* patients with ≥ grade 2 pre-existing peripheral neuropathy, history of allergic reactions to the chemotherapeutic agents, and uncontrolled intercurrent diseases as well as HIV positive patients.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
locoregional recurrence free survival in months | 1 years
  comparison of the locoregional recurence free survival in both arms

SECONDARY OUTCOMES:
overall survival | 5 years
  overall survival in months in both arms

CONTACTS AND LOCATIONS:
Overall Officials: doAA ABDELALEEM, Master, Principal Investigator — Assiut University

REFERENCES:
- See also: Concurrent chemotherapy and radiotherapy for organ preservation in advanced larynx cancer. N Engl J Med. 2003; 349:2091-2098. — https://www.ncbi.nlm.nih.gov/pmc/articles/pmc3577950/